CLINICAL TRIAL: NCT01779323
Title: Prospective Study of Urethral Mobility in Male Stress Urinary Incontinence Pre- and Post- Placement of Transobturator Sling
Brief Title: Study of Urethral Mobility in Male Stress Urinary Incontinence Pre- and Post- Placement of Transobturator Sling
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00026977
Record Dates: First submitted 2013-01-28; First posted 2013-01-30 (Estimated); Last update posted 2023-08-16 (Actual); Status verified 2016-03

CONDITIONS: Male Stress Urinary Incontinence
Keywords: SUI; stress urinary incontinence; male; transobturator sling
MeSH Terms: conditions — Urinary Incontinence, Stress | interventions — Lead

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pre and Post Sling Pelvic MRI: Cohort: Measure change in hypermobility of urethra after transobturator sling surgery via pelvic MRI.
  Interventions: Other: Pre and Post Sling Pelvic MRI

INTERVENTIONS:
Other: Pre and Post Sling Pelvic MRI — Pre and Post Sling Pelvic MRI
  Other Names: Transobturator suspension sling system (TOS), AMS Advance

SUMMARY:
The hypothesis is men with stress urinary incontinence, including those following radical retropubic prostatectomy and other prostate surgery, have preoperative urethral mobility as measured by magnetic resonance imaging (MRI) that improves significantly following sling placement. The investigators theorize that the sling helps with primary hypermobility of this pathophysiologic cause of stress urinary incontinence.

ELIGIBILITY:
Inclusion Criteria:

* The control group:
* normal male subjects
* The Intervention group:
* male
* with stress urinary incontinence
* 45 years or older
* history of prior radical prostatectomy
* complains of stress urinary incontinence
* scheduled for a transobturator sling surgery
* ability and willingness to provide written consent

Exclusion Criteria:

* absolute or relative contraindications to MRI
* claustrophobia
* inability to undergo the male sling surgery
* PI judgement

Absolute contraindications to MRI:

* electronically, magnetically, and mechanically activated implants
* ferromagnetic or electronically operated active devices
* metallic splinters in the eye
* ferromagnetic hemostatic clips in the central nervous system

Relative contraindications to MRI:

* cochlear implants
* other pacemakers
* nerve stimulators
* lead wires or similar wires
* prosthetic heart valves
* hemostatic clips
* non-ferromagnetic stapedial implants

Min Age: 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients from the urology clinic.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2012-03; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Change in urethral mobility | Within 2-5 months after enrollment
  Measure change in urethral mobility from baseline versus 2-5 months post-surgery versus no surgical intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Peterson, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States